CLINICAL TRIAL: NCT01872325
Title: Improving the Cardiac Arrest Diagnostic Accuracy of 9-1-1 Emergency Medical Dispatchers
Brief Title: Improving Cardiac Arrest Diagnostic Accuracy of Emergency Medical Dispatchers
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0379-01H
Record Dates: First submitted 2013-05-09; First posted 2013-06-07 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; bystander cardiopulmonary resuscitation CPR; dispatch-assisted CPR instructions; agonal breathing
MeSH Terms: conditions — Heart Arrest | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Training site: All emergency medical dispatchers at a central ambulance communication centre in Ontario will participate in an educational program designed to improve cardiac arrest diagnostic accuracy.
  Interventions: Behavioral: Education
- Control site: All emergency medical dispatchers at a central ambulance communications centre geographically remote from the Training Site and has a similar rate to the Training Site for cardiac arrests, bystander CPR rate, and survival

INTERVENTIONS:
Behavioral: Education — An education program will be developed using behaviour change techniques specifically mapped to address modifiable factors identified in a previous study. These techniques will include: information about the significance of agonal breathing, modeling/demonstration of desired behavioural skills, rehearsal of desired skills, and monitoring/reinforcement and feedback.
  Groups: Training site

SUMMARY:
The main goal of this project is to help 9-1-1 emergency medical dispatchers save the lives of more cardiac arrest victims. The investigators will develop teaching tools to help the dispatchers recognize abnormal breathing that may indicate a victim as having a cardiac arrest. After training sessions, the investigators will see if dispatchers can get better at recognizing abnormal breathing, how often they give CPR instructions, and if use of the teaching tool will increase bystander CPR and the number of victims leaving the hospital alive.

DETAILED DESCRIPTION:
Cardiac arrest is a leading cause of death in Canada; it is defined as the sudden cessation of cardiac mechanical activity. It is uniformly fatal if not treated within minutes. More than 85% of out-of-hospital cardiac arrest (OOHCA) occur in residential locations so public access to automatic external defibrillators, to restart the heart, are not helpful. The overall rate of survival for OOHCA rarely exceeds 8%.

Bystander cardiopulmonary resuscitation (CPR) is chest compression and ventilations provided by someone not on the emergency response team. A victim or cardiac arrest is almost 4 times more likely to survive when receiving bystander CPR. However, despite various attempts to improve bystander rates they have remained low, not exceeding 15% in Ontario. It has been shown that since the ambulance dispatch centres in Ontario implemented dispatch-assisted CPR instructions (given to callers while emergency vehicles were on the way), there was a significant increase in use.

Emergency medical dispatchers can identify about 70% of OOHCA cases over the phone. Agonal breathing (laboured breathing preceding death) may be misinterpreted as a sign of life, and is responsible for as much as 50% of missed diagnoses. There is no specific training on the significance of this sign, and minimal information about recognizing cardiac arrest. An educational intervention designed to better understand the significance of agonal breathing and to clarify the existing CPR instruction protocol will most likely increase the frequency of CPR instructions, bystander CPR rates, and potentially survival of victims of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* presumed cardiac origin
* event occurs in the catchment area of Training or Control Site
* resuscitation is attempted by a bystander and/or the emergency responders

Exclusion Criteria:

* patients younger than 16 years old
* patients who are "obviously dead" as defined by the Ambulance Act of Ontario (decomposition, rigor mortis, decapitation, or other)
* trauma victims including hanging and burns
* cardiac arrest of non-cardiac origin including drug overdose, carbon monoxide poisoning, drowning, exsanguination, electrocution, asphyxia, hypoxia related to respiratory disease, cerebrovascular accident, and documented terminal illness

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with out-of-hospital cardiac arrest
Sampling Method: Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD,MSc,FRCPC, Principal Investigator — The Ottawa Hospital Research Institute and University of Ottawa
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Training Site | Control Site
Started | 689 | 387
Completed | 689 | 387
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training Site | Control Site | Total
Number analyzed (Participants) | 689 | 387 | 1076
Age, Continuous [Mean (Full Range); unit: years] | 68 [16 to 100] | 68 [22 to 98] | 68 [16 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 136 | 353
  Male | 472 | 251 | 723
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 689 | 387 | 1076
Witnessed Status [Count of Participants; unit: Participants] — A witnessed cardiac arrest is seen or heard by someone other than Emergency Medical Services (lay person, a healthcare provider, a police officer or an off-duty fire/Emergency Medical Services provider who is not part of the organized response).
  Participants | 310 | 162 | 472
Initial Cardiac Rhythm Ventricular Fibrillation/Ventricular Tachycardia [Count of Participants; unit: Participants] | 199 | 87 | 286

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Agonal Breathing
Description: By reviewing recordings of all cardiac arrest calls, including missed cases retrieved from a registry, document presence or absence of agonal breathing.
Time Frame: At the time of the cardiac arrest event
Measure: Count of Participants; unit: Participants
Arm/Group | Training Site | Control Site
Number analyzed (Participants) | 689 | 387
Participants | 176 | 87

2. Secondary Outcome: Number of Cases Where Cardiac Arrest Was Recognized by the Ambulance Dispatcher
Description: By reviewing recordings of all cardiac arrest calls, collect information on dispatcher recognition of cardiac arrest to bystander implementation of chest compressions
Time Frame: At the time of the cardiac arrest event
Measure: Count of Participants; unit: Participants
Arm/Group | Training Site | Control Site
Number analyzed (Participants) | 689 | 387
Participants | 495 | 287

3. Other Pre Specified Outcome: Number of Participants Who Received Bystander CPR
Description: The first member of the emergency response team to arrive at scene will document whether or not chest compressions have been initiated by someone prior to the arrival of emergency team
Time Frame: At the time of the cardiac arrest event
Measure: Count of Participants; unit: Participants
Arm/Group | Training Site | Control Site
Number analyzed (Participants) | 689 | 387
Participants | 247 | 153

4. Other Pre Specified Outcome: Number of Participants Surviving to Hospital Discharge
Description: Accessing hospital medical records or coroner's reports, assess survival of cardiac arrest victim as being discharged alive from hospital
Time Frame: At the time of the cardiac arrest event to discharge alive from hospital (varies, depending on length of hospital stay)
Measure: Count of Participants; unit: Participants
Arm/Group | Training Site | Control Site
Number analyzed (Participants) | 689 | 387
Participants | 86 | 27

ADVERSE EVENTS:
Arm/Group | Training Site | Control Site
Serious Adverse Events (participants affected / at risk) | 0/689 | 0/387
Other Adverse Events (participants affected / at risk) | 0/689 | 0/387

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No